CLINICAL TRIAL: NCT07235228
Title: Effects of Vivatlac Synbiotic on the Gut Microbiota of Patients With Irritable Bowel Syndrome - A Randomized, Double-blind, Placebo-Controlled, 12 Weeks Clinical Trial
Brief Title: Effects of Vivatlac Synbiotic on Gut Micribiota of IBS Patients
Acronym: ViIBS3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kalisz 2025-02 ViIBS Trial III
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; Vivatlac synbiotic; synbiotic; ViIBS III trial; gut microbiota; 16S rRNA sequencing; nanopore shotgun sequencing; Clostridioides difficile; fecal calprotectin; gut inflammation
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized allocation of IBS patients to a synbiotic or a placebo group of similar size
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Capsule containing maize starch with identical appearance as verum. One capsule taken per day before bedtime. Treatment duration 12 weeks.
  Interventions: Dietary Supplement: Placebo
- Vivatlac Synbiotic (Experimental): Vivatlac Synbiotic for 12 weeks. One capsule containing a mixture of nine different probiotic bacteria with a total amount of 4.5 x 10^9 colony forming units and 63 mg of fructooligosaccharides. One capsule taken per day before bedtime. Treatment duration 12 weeks.
  Interventions: Dietary Supplement: Vivatlac Synbiotic

INTERVENTIONS:
Dietary Supplement: Vivatlac Synbiotic — Vivatlac Synbiotic containing a total of 4.5 x 10^9 colony forming units (CFU) of nine different probiotic bacteria. Probiotic bacteria strains and their CFU amount per capsule are: Lactococcus lactis Ll-23, 9.00 x 10^8 CFU; Lactobacillus helveticus SP 27, 9.00 x 10^8 CFU; Bifidobacterium longum Bl-05, 6.75 x 10^8 CFU; Bifidobacterium longum ES1, 4.50 x 10^8 CFU; Lacticaseibacillus rhamnosus Lr-32, 4.50 x 10^8 CFU; Streptococcus thermophiles St-21, 4.50 x 10^8 CFU; Lacticaseibacillus casei Lc-11, 2.25 x 10^8 CFU; Lactiplantibacillus plantarum Lp-115, 2.25 x 10^8 CFU; Bifidobacterium bifidum Bb-02, 2.25 x 10^8 CFU. As a prebiotic component each capsule contains 63 mg of fructooligosaccharides.
  Arms: Vivatlac Synbiotic
Dietary Supplement: Placebo — Capsule containing maize starch with identical appearance as verum.
  Arms: Placebo

SUMMARY:
Multi-center, randomized, double-blind, placebo-controlled, 12 weeks trial investigating the effects of a nine-strain synbiotic (Vivatlac Synbiotikum) on the gut microbiota of IBS patients

DETAILED DESCRIPTION:
The study design is a multi-centre, randomized, double-blind, placebo-controlled clinical trial in patients diagnosed with Irritable Bowel Syndrome (IBS). Diagnosis of IBS is performed with the World Gastroenterology Organisation's IBS questionnaire for health care providers. Assessment of the severity of IBS is done by using the IBS Severity Scoring System (IBS-SSS). IBS patients with moderate to severe IBS will be included in the study (IBS-SSS ≥ 175). A four-week treatment-free screening phase is used to evaluate the patients' IBS symptoms and stool characteristics using a patient diary.

The screening phase is followed by treatment with one capsule per day of a nine-strain synbiotic (Vivatlac® Synbiotikum) or with an identical-looking placebo for twelve weeks.

Each capsule of Vivatlac® Synbiotikum contains a total of 4.5 x 10^9 colony-forming units (CFU) of nine different probiotic bacteria. Probiotic bacteria strains and their CFU amount per capsule are: Lactococcus lactis Ll-23, 9.00 x 10^8 CFU; Lactobacillus helveticus SP 27, 9.00 x 10^8 CFU; Bifidobacterium longum Bl-05, 6.75 x 10^8 CFU; Bifidobacterium longum ES-1, 4.50 x 10^8 CFU; Lacticaseibacillus rhamnosus Lr-32, 4.50 x 10^8 CFU; Streptococcus thermophiles St-21, 4.50 x 10^8 CFU; Lacticaseibacillus casei Lc-11, 2.25 x 10^8 CFU; Lactiplantibacillus plantarum Lp-115, 2.25 x 10^8 CFU; Bifidobacterium bifidum Bb-02, 2.25 x 10^8 CFU. In addition, each capsule contains 68 mg of fructooligosaccharides (FOS).

Treatment effects on severity of IBS symptoms is assessed by using the IBS-Severity Scoring System (IBS-SSS), before the start of treatment and after 4, 8, and 12 weeks of treatment. Changes of IBS severity is assessed by using the IBS-Global Improvement Scale (IBS-GIS), before the start of treatment and after 4, 8, and 12 weeks of treatment. Patients are assessed for IBS adequate relief by using the IBS-Adequate Relief scale (IBS-AR), after 4, 8, and 12 weeks of treatment. Stool form characteristics is assessed with the Bristol Stool Form Scale (BSFS), at the start of the screening phase, at the start of treatment, and after 4, 8, and 12 weeks of treatment.

Stool samples are taken from all patients before the start of treatment and after 12 weeks of treatment. Fecal samples will be analyzed for gut microbiota profiles using 16S rRNA sequencing (taxonomic identification of bacterial genera) and/or nanopore shotgun sequencing (species-level identification). The presence of gut inflammation will be assessed by measuring fecal calprotectin as a biomarker for gut inflammation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for Irritable Bowel Syndrome using the IBS questionnaire for Health Care Providers of the World Global Gastroenterology Organization
* IBS severity assessed with the IBS-Severity Scoring System (IBS-SSS) being ≥ 175 points (indicating medium or severe IBS).

Exclusion Criteria:

* patients currently taking products containing probiotics or have taken this kind of products during the last 3 months
* patients currently taking antibiotics or have taken antibiotics during the last 3 months
* patients having a concurrent severe illness (malignancies, uncontrolled hypertension or diabetes, hepatic, renal or cardiac dysfunctions, serious neurological disorders, psychosis, respiratory disorders such as asthma or COPD, hyper- or hypothyroidism
* patients having chronic bowel disorders other than IBS, including inflammatory bowel disease, gastroenteritis, stomach and duodenal cancer, celiac disease
* patient being tested positive for presence of Clostridioides difficile
* patient being pregnant, lactating, or planning to become pregnant during the next 3 months
* patient being diagnosed to have a lactose intolerance
* patients using motility drugs or dietary fiber supplements withing 2 weeks before study start
* patient taking anti-coagulant medication
* patients have participated in another clinical trial within the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of gut-microbiota composition using 16S rRNA sequencing (taxonomic identification of bacterial genera) | Measured before the start of treatment and at the end of the 12-week treatment.
  Fecal samples are collected from patients and frozen as quickly as possible at -20 °C until further analysis. Samples are analyzed by 16S rRNA sequencing for a taxonomic identification of bacterial genera. Sample compositions are compared between placebo and synbiotic group before the start of the treatment and after 12 weeks of treatment.
Changes of gut-microbiota composition using nanopore shotgun sequencing (species-level identification) | Measured before the start of treatment and at the end of the 12-week treatment
  Fecal samples are collected from patients and frozen as quickly as possible at -20 °C until further analysis. Samples are analyzed by nanopore shotgun sequencing for a species level identification of bacterial genera. Sample compositions are compared between placebo and synbiotic group before the start of the treatment and after 12 weeks of treatment.

SECONDARY OUTCOMES:
Measurement of calprotectin levels in fecal samples | Measured before the start of treatment and at the end of the 12-week treatment.
  Fecal samples are collected from patients and frozen as quickly as possible at -20 °C until further analysis. Samples are frozen as fast as possible at minus 20°C. Stool samples are stored at minus 20°C until further processing. Single-use Calex® Caps (Bühlmann Laboratories, Schönenbuch, Switzerland) are used according to the manufacturer's instructions to prepare samples for measurements. Calprotectin concentrations are determined using the QB® fCAL extended test (Bühlmann Laboratories, Schönenbuch, Switzerland) in combination with a Quantum Blue® Reader II BI-POCTR-ABS (Bühlmann Laboratories, Schönenbuch, Switzerland). The difference in the fecal Calprotectin concentration in stool samples taken from patients of the placebo and the synbiotic group are compared.
Severity of IBS using the IBS-Severity Scoring System (IBS-SSS) | Measured at enrollment, start of the treatment phase, and after 4, 8, and 12 weeks of treatment.
  IBS-Severity Scoring System is a 5-question survey that asks: 1. the severity of abdominal pain, 2. frequency of abdominal pain, 3. severity of abdominal distention, 4.dissatisfaction with bowel habit, and 5. interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Each of the five question generates a maximum score of 100 point, and total scores can range from 0-500 with higher scores indicating severe symptoms. A decrease of 50 points is associated with a clinically meaningful improvement.
Changes of IBS severity using the IBS Global Improvement Scale (IBS-GIS) | Measured at the start of the treatment phase, and after 4, 8, and 12 weeks of treatment.
  Patients answer the question "Have you felt any change in the severity of your symptoms over the past 7 days compared to how you felt before the medicine was given?
  The answers are recorded based on the 7-point scale:
  * I feel that the symptoms have worsened significantly (1 point)
  * I feel that the symptoms have moderately worsened (2 points)
  * I feel that the symptoms have slightly worsened (3 points)
  * I feel no change (4 points)
  * I feel a slight improvement (5 points)
  * I feel moderate improvement (6 points)
  * I feel significant improvement (7 point) IBS-GIS score indicates: improvement if is >4 or worsening if is<4, no change if is 4
Changes in adequate relief of IBS-symptoms (IBS-AR) | Measured at the start of the treatment phase, and after 4, 8, and 12 weeks of treatment.
  The IBS-Adequate Relief (IBS-AR) scale is a dichotomous single item scale that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms? The answer is YES or NO.
Changes of stool form characteristics with the Bristol Stool Form Scale (BSFS) | Measured at the start of the treatment phase, and after 4, 8, and 12 weeks of treatment.
  The type of stool is assessed using the Bristol Stool Form Scale (BSFS). Pateint have to select from seven stool pictures the picture ressembling the most their own stool form. The BSFS is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Piatek, Prof. Dr., Principal Investigator — The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz
Locations (1):
- State Hospital Jarocin, Jarocin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piatek J, Krauss H, Ciechelska-Rybarczyk A, Bernatek M, Wojtyla-Buciora P, Sommermeyer H. In-Vitro Growth Inhibition of Bacterial Pathogens by Probiotics and a Synbiotic: Product Composition Matters. Int J Environ Res Public Health. 2020 May 11;17(9):3332. doi: 10.3390/ijerph17093332. PMID 32403297
- [Background] Sommermeyer H, Pituch HM, Wultanska D, Wojtyla-Buciora P, Piatek J, Bernatek M. Inhibition of Quinolone- and Multi-Drug-Resistant Clostridioides Difficile Strains by Multi Strain Synbiotics-An Option for Diarrhea Management in Nursing Facilities. Int J Environ Res Public Health. 2021 May 30;18(11):5871. doi: 10.3390/ijerph18115871. PMID 34070727
- [Background] Piatek J, Sommermeyer H, Bernatek M, Ciechelska-Rybarczyk A, Oleskow B, Mikkelsen LS, Barken KB. Persistent infection by Salmonella enterica servovar Typhimurium: are synbiotics a therapeutic option? - a case report. Benef Microbes. 2019 Mar 13;10(2):211-217. doi: 10.3920/BM2018.0080. Epub 2018 Dec 21. PMID 30574800
- [Background] Sommermeyer H, Piatek J. Synbiotics as Treatment for Irritable Bowel Syndrome: A Review. Microorganisms. 2024 Jul 21;12(7):1493. doi: 10.3390/microorganisms12071493. PMID 39065261
- [Background] Sommermeyer H, Chmielowiec K, Bernatek M, Olszewski P, Kopczynski J, Piatek J. Results from a Cross-Sectional Observational Study Examining Irritable Bowel Syndrome Patients Six Months After Finishing Their Participation in the ViIBS Trial. Nutrients. 2024 Nov 15;16(22):3911. doi: 10.3390/nu16223911. PMID 39599697
- [Background] Sommermeyer H, Chmielowiec K, Bernatek M, Olszewski P, Kopczynski J, Piatek J. Effectiveness of a Balanced Nine-Strain Synbiotic in Primary-Care Irritable Bowel Syndrome Patients-A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2024 May 16;16(10):1503. doi: 10.3390/nu16101503. PMID 38794741